CLINICAL TRIAL: NCT03637998
Title: The Impact of Physical Activity on the Neurophysiologic and Gene Expression Profiles of Chronic Low Back Pain: A Longitudinal Study Protocol
Brief Title: Physical Activity on Neurophysiologic Gene Expression Profiles of Chronic Low Back Pain
Acronym: PROPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wanli Xu, Assistant Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-086; 5P20NR016605 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low Back Pain; Self-Management
Keywords: Gene expression; Quantitative Sensory Testing; Genotyping
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROPEL (Experimental): The Problem-solving Pain to Enhance Living Well (PROPEL) intervention entails each participant watching 10 video modules via REDCap. These modules include: (1) pain neurophysiology, (2) catastrophizing, (3) stress reactivity, (4) fear of movement, (5) progressive relaxation, (6) deep breathing, (7) guided imagery, (8) heat, ice and stretching, (9) strategies for physical activity self-activation and (10) problem-solving.
  Interventions: Behavioral: Problem-solving Pain to Enhance Living Well (PROPEL)

INTERVENTIONS:
Behavioral: Problem-solving Pain to Enhance Living Well (PROPEL) — PROPEL incorporates evidence-based, standard of care methods to promote physical activity among individuals with pain, and tools to improve knowledge, skills and confidence to cope with cLBP. The focus is self-management of cLBP. All eligible participants will then undergo baseline data collection, which entails completion of study questionnaires, quantitative sensory testing (QST) and venipuncture for collection of a blood specimen. Participants will be provided with the information to access the PROPEL intervention. All participants will be asked to complete questionnaires at 2, 4, 6, 8, and 10 weeks following baseline testing. At 12 weeks, participants will be scheduled for a final data collection visit, which will follow the same procedures as the baseline visit.

SUMMARY:
This pilot project will provide an understanding of the contextual variables responsible for chronic low back pain. These variables include, genetic variation, pain sensitivity, reactivity, pain catastrophizing, perceived stress and kinesiphobia. The purpose is to understand the initial efficacy of self-management (SM) strategies on each of these contextual variables, in an effort to inform a personalized approach to managing chronic low back pain and its effect on improved health outcomes.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is the second most frequent chronic pain condition in the United States and results in billions of dollars each year in health care expenses, disability and lost productivity. A major factor that contributes to the refractory nature of cLBP is enhanced pain sensitivity, which is an altered state of pain processing that amplifies pain sensation and impairs descending pain inhibition. Enhanced pain sensitivity in patients who develop cLBP is associated with altered expression of pro-nociceptive and inflammatory genes. On the other hand, regular physical activity of at least moderate intensity for 150 or more minutes per week is recommended to reduce pain severity and improve function in individuals with cLBP. Therefore, a deeper mechanistic understanding of the effect of physical activity on the neurophysiologic and gene transcription alterations that characterize cLBP may inform more specific treatment options to optimize pain reduction and reduce the risk of pain chronicity.

The purpose of this longitudinal cohort pilot study is to examine the feasibility, acceptability, and preliminary efficacy of the Problem-solving Pain to Enhance Living Well (PROPEL) self-management (SM) intervention on cLBP. This pre-post intervention study will recruit 40 community dwelling adults (age 18 - 60 years old) with cLBP. They will receive electronic video modules focused on cLBP SM knowledge and weekly phone consultations to facilitate monitoring and problem-solving. All participants will be assessed for primary outcomes including cLBP SM behaviors, physical activity, pain severity and interferance, and pain sensitivity at baseline and every 2 weeks for 12 weeks. The study will examine differential neurophysiologic and gene expression profiles between participants with cLBP at 12-weeks post-intervention and correlate these outcome measures to total duration of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* be 18-60 years of age;
* have nonspecific cLBP (≥4 on the numeric rating scale; NRS) present for at least 3 out of the last 6 months and ≥ half the days in the past 6 months;
* comprehend English (due to lack of reliability and validity of study instruments and the intervention in non-English populations).
* Have daily access to a computer, tablet or smartphone with access to internet
* Have less than 150 minutes of moderate physical activity a week
* Be willing to wear activity tracker for 12 weeks

Exclusion Criteria:

* Chronic pain at another site or associated with a painful condition (eg., fibromyalgia, neuropathy, rheumatoid arthritis)
* history of comorbidities that affect sensorimotor function (eg., multiple sclerosis, cancer, spinal cord injury, diabetes)
* previous spinal surgery within last 1 year
* presence of neurological deficits such as weakness in the lower extremities (motor strength 4/5 of quads, glutes, hamstrings, EHL)
* bowel or bladder dysfunction such as difficulty voiding or incontinence
* sciatica or (+) leg raise
* positive Romberg test
* being pregnant or within 3 months postpartum
* history of psychological disorders (major depression, bipolar disorder, schizophrenia)
* identification of any "red flag" condition in the volunteer's past medical history that suggests specific LBP as determined by Dr. Kim such as conditions or medications that can affect pain sensitivity
* injury to non-dominant hand or presence of open skin lesions, disturbed sensation, carpal tunnel or rash

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Baseline, 2, 4, 6, 8, 10 and 12 weeks
  Fitbit for activity tracker

SECONDARY OUTCOMES:
Change in gene expression profiles | Baseline and 12 weeks post-intervention
  RNA sequencing
Change in pain sensitivity | Baseline and 12 weeks post-intervention
  Quantitative sensory testing
Relationship between pain self-management and pain severity | Baseline, 2, 4, 6, 8, 10 and 12 weeks
  Change over time through questionnaires
Relationship between pain self-management and pain interferance | Baseline, 2, 4, 6, 8, 10 and 12 weeks
  Change over time through questionnaires
Relationship between pain self-management and quality of life | Baseline, 2, 4, 6, 8, 10 and 12 weeks
  Change over time through questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wanli Xu, PhD, Principal Investigator — University of Connecticut; Angela Starkweather, PhD, Study Director — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that are part of National Institute of Nursing Research (NINR) designated common data elements collected during the trial, after de-identification have been submitted to NIH repository at the Common Data Repository for Nursing Science (cdRNS). Data can be accessed by directly submitting requests at that website.
  When will data be available (start and end dates)? Immediately. No end date.
  With whom? Anyone who wishes to access the data and creates an account on cdRNS.nih.gov.
  By what mechanism will data be made available? Data are available at cdRNS.nih.gov
Time Frame: Within 2 years
Access Criteria: Requests will be submitted through the cdRNS website
URL: https://cdrns.nih.gov

REFERENCES:
- [Derived] Xu W, Zhang Y, Wang Z, Dorsey SG, Starkweather A, Kim K. Pain self-management plus activity tracking and nurse-led support in adults with chronic low back pain: feasibility and acceptability of the problem-solving pain to enhance living well (PROPEL) intervention. BMC Nurs. 2023 Jun 25;22(1):217. doi: 10.1186/s12912-023-01365-y. PMID 37355622
- See also: Center for Accelerating Precision Pain Self-Management (CAPPS-M) Website — https://cappsm.nursing.uconn.edu/